CLINICAL TRIAL: NCT07093346
Title: The Impact of Pectin Supplementation on Systematic Inflammation Pathway, Gut Microbiome, and Metabolic Health in Patients With Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD): A Randomised, Placebo-Controlled, Dietary Intervention Study
Brief Title: The Impact of Pectin Supplementation on Systematic Inflammation Pathway, Gut Microbiome, and Metabolic Health in Patients With Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Acronym: PEC-MASLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 24076; 351797 (Other: IRAS)
Record Dates: First submitted 2025-07-08; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-04

CONDITIONS: Nonalcoholic Fatty Liver Disease; Nonalcoholic Fatty Liver Disease (NAFLD); MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; MASLD; NAFLD; Metabolic Dysfunction-Associated Steatotic Liver Disease; NAFLD (Nonalcoholic Fatty Liver Disease); NAFLD (Non-alcoholic Fatty Liver Disease); NAFLD - Non-Alcoholic Fatty Liver Disease; NAFLD - Nonalcoholic Fatty Liver Disease
Keywords: LM pectin; pectin; MASLD; NAFLD; Nonalcoholic Fatty Liver Disease; Systemic Inflammatory Response; Dietary Fiber; Dietary Fibre; Diet; gut microbiota; Metabolic Dysfunction-Associated Steatotic Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Pectins; Chocolate; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: The study will be a parallel design, placebo-controlled, randomised dietary intervention study in which each participant will be randomly assigned to either pectin supplementation arm or control arm using online software (sealedenvelope.com).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pectin (Active Comparator): 15g/day of pectin with 10g/day of cocoa powder added as flavour will be provided to participants for 6 weeks.
  Interventions: Dietary Supplement: Pectin
- Cocoa Powder (Placebo Comparator): 10g/day of cocoa powder will be provided to participants for 6 weeks.
  Interventions: Other: Cocoa Powder
- Magnetic resonance imaging (MRI) Validation (Other): To validate MRI scans as a tool to assess intestinal wall thickness to indicate gut permeability on MASLD patients, the investigators will scan 15 healthy volunteers twice, at baseline and after 6 weeks, and then compare their results with MASLD participant results at baseline and after 6 weeks.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging with Contrast

INTERVENTIONS:
Dietary Supplement: Pectin — 15g of pectin with 10g of cocoa powder added as flavour were randomly allocated to eligible participants.
  Arms: Pectin
Other: Cocoa Powder — 10g of cocoa powder served as the control/ placebo to compare the effects observed with pectin.
  Arms: Cocoa Powder
Diagnostic Test: Magnetic Resonance Imaging with Contrast — To validate MRI scans as a tool to assess intestinal wall thickness to indicate gut permeability on MASLD patients, the investigators will scan 15 healthy volunteers twice, at baseline and after 6 weeks, and then compare their results with MASLD participant results at baseline and after 6 weeks.
  Other Names: MRI
  Arms: Magnetic resonance imaging (MRI) Validation

SUMMARY:
The goal of this clinical trial is to learn if daily supplementation with Low-methoxy (LM) pectin (polysaccharides extracted from citrus peels), which are commonly found in the UK diet (not pharmacological agents), can reduce systemic inflammation and improve gut microbiota composition in adults recently diagnosed with Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD). The main question it aims to answer is:

-How does dietary Low-methoxy (LM) pectin supplementation affect systematic inflammation pathways such as those mediated by gut microbiota composition and what are the impacts on general metabolic indicators in individuals with MASLD?

Researchers will compare a group taking 15g of LM-pectin with 10g of cocoa powder to a placebo group receiving 10g of placebo with 10g of cocoa powder to see if LM-pectin has measurable effects on inflammation and gut microbiota.

Participants will:

* Take a daily supplement for 6 weeks: either 15g of LM-pectin with 10g of cocoa powder (intervention), or 10g of placebo with 10g of cocoa powder (control)
* Provide stool and fasting blood samples before and after the intervention
* Undergo anthropometric measurements (weight, height, waist/hip ratio, and blood pressure)
* Complete a case report form (CRF) including demographics and health/medical history
* Undergo a FibroScan™ to assess liver health
* (Optional) Participate in MRI scans to evaluate gut permeability

DETAILED DESCRIPTION:
Primary Objective:

This research aims to study the effects of daily ingestion of LM pectin on inflammation pathways by measuring the blood inflammatory markers associated with physiological processes (TNFα, IL-6, IL-10, IFNᵞ, C - reactive protein, Zonulin (Haptoglobulin), IL-1β).

Secondary Objectives:

1. Assessment of changes in anthropometric measures.
2. Assessment of changes in general metabolic indicators, such as fasting blood glucose and other blood-based markers relevant to MASLD (e.g., CK18-M30, CK18-M65, PROC3, Enhanced Liver Fibrosis (ELF), NIS2+™, YKL-40, microRNA miR-34a-5p, liver-associated enzymes such as Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), gamma-glutamyl transferase (GGT), Alkaline Phosphatase (ALP)), bilirubin levels, lipid profiles, and platelet counts.
3. Exploration of changes in gut microbiome composition.
4. Exploration of modifications in non-invasive physiological assessments linked to liver characteristics, such as fat content and stiffness through controlled attenuation parameter (CAP) and transient elastography.
5. Observation of alteration in fat in liver and other surrounding abdominal organs through Dixon MRI sequence in patients who will agree to have 2 MRI scans.
6. Validation of MRI measures (T2*) as a tool to measure gut permeability among MASLD patients and investigation of changes in gut permeability in participants undergoing two MRI scans.
7. Investigation the presence of gene variants such as MUC2, encoding Mucin protein, that are associated with gut permeability.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the main study:

* Patients with clinical diagnosis of MASLD (formerly termed non-alcoholic fatty liver disease (NAFLD)), having assessment suggesting that liver fat > 5% (e.g. histological evidence or/ and Transient Elastography using Controlled Attenuation Parameter (CAP)- FibroScan™ in the past month and/or liver imaging (such as ultrasound, computerized tomography (CT) or magnetic resonance imaging (MRI)).
* Participants willing and able to give informed consent for participation in the study.
* Participants aged ≥18 years who have a body mass index (BMI) between 18.5 and 39.9 kg/m2 and stable weight (weight gain or loss ≤ 3kg) for the past 3 months.
* For diabetic participants: controlled blood glucose levels Haemoglobin A1C (HbA1c) <7.0% (<53 mmol/mol) [1].
* Able to undergo CAP-FibroScan™.

Inclusion criteria for healthy participants who will have MRI scans:

* Participants willing and able to give informed consent for participation in the study.
* Participants aged ≥18 years.
* participants with CAP<250 kpa<8kP by a FibroScan™ within the past 6 months.

Exclusion Criteria:

Exclusion criteria for the main study:

* Have allergy toward soya, milk or chocolate.
* Have allergy toward pectin.
* Participants on vegan diet.
* Have eating disorders or difficulties or gastrointestinal conditions e.g. malabsorptive conditions such as coeliac, Irritable Bowel Syndrome (IBS) or Inflammatory Bowel Disease (IBD) or gastroparesis.
* Have chronic malnutrition condition.
* History of major surgery which potentially limits participation or completion of the study.
* History of previous intestinal surgery known to affect food intake or digestive function, including bariatric surgery.
* Use of antibiotics, antifungal medications, probiotics or prebiotics 90 days before the start of the study.
* Are taking the following medications: immunosuppressants, amiodarone and/or perhexiline.
* Are currently following or anticipated to commence a specialised commercially available weight loss diet and/or program or concomitant use of any weight loss medication or herbal weight loss products.
* History of side effects towards probiotics or prebiotics.
* History or current psychiatric illness.
* History or current neurological condition (e.g. epilepsy).
* Participants with other liver abnormalities.
* Evidence of monogenic metabolism diseases such as Lysosomal acid lipase deficiency (LALD), Wilson disease, Hypobetalipoproteinemia, or inborn errors of metabolism.
* Have had a weight change exceeding 3 kg within 3 months.
* Uncontrolled diabetes, active malignancy, or chronic infections.
* Having symptoms of active infection.
* Excessive alcohol intake defined as self-reported intakes greater than 21 units per week in men, and 14 units per week in women.
* Participants who are pregnant, breast feeding or actively planning pregnancy will be excluded from the study.
* Participation in any other trial in the last 3 months.

Exclusion criteria for healthy volunteers MRI scans and patients optional MRI scans:

* Contraindications for MRI scanning: having pacemakers, defibrillators, neurostimulators, prohibited medical implants, and foreign bodies (e.g. bullets, shrapnel, metal slivers), history of metallic foreign body in eye(s) and penetrating eye injury that could present a risk during an MRI scan.
* Difficulty breathing or inability to lie flat, as well as conditions that could worsen under stress (such as anxiety or panic disorders, claustrophobia, uncontrolled hypertension, or seizure disorders) severe enough to prevent undergoing an MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of blood markers contributing to systemic inflammation pathway (TNFα (pg/mL), IL-6 (pg/mL), IL-10 (pg/mL), IFNᵞ (pg/mL), C-Reactive Protein (pg/mL), Zonulin (Haptoglobulin)(pg/m), IL-1β(pg/mL)). | 6 weeks
  Change in circulating markers of inflammation measured by ELISAs in serum samples collected pre and post the 6-weeks intervention period.

SECONDARY OUTCOMES:
Change in BMI (kg/m²) | 6 weeks
  Changes in BMI pre and post the 6-weeks intervention period.
Assessment of changes in general metabolic indicators, such as fasting blood glucose and other blood-based markers relevant to MASLD (e.g., CK18-M30, CK18-M65, PROC3, Enhanced Liver Fibrosis (ELF), NIS2+™, YKL-40, microRNA miR-34a-5p) | 6 weeks
  Changes in general metabolic indicators, such as fasting blood glucose and other blood-based markers relevant to MASLD (e.g., CK18-M30, CK18-M65, PROC3, Enhanced Liver Fibrosis (ELF), NIS2+™, YKL-40, microRNA miR-34a-5p) pre and post the 6-weeks intervention period.
Assessment of changes in liver-associated enzymes such as Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), gamma-glutamyl transferase (GGT), Alkaline Phosphatase (ALP)), bilirubin levels, lipid profiles, and platelet counts. | 6 weeks
  Changes in liver-associated enzymes such as Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), gamma-glutamyl transferase (GGT), Alkaline Phosphatase (ALP)), bilirubin levels, lipid profiles, and platelet counts pre and post the 6-weeks intervention period.
Change in Liver Stiffness via Transient Elastography | 6 weeks
  CAP and liver stiffness (in kPa) measured using transient elastography.
Change in Liver Fat Fraction Assessed by Dixon MRI Sequence. | 6 weeks
  Fat fraction (%) in liver and abdominal organs assessed using Dixon MRI before and after the 6-week intervention.
Change in Intestinal Permeability Measured by T2* MRI. | 6 weeks
  T2* values in gut wall tissue will be compared before and after the intervention as a proxy for gut permeability.
Investigation the presence of gene variants such as MUC2, encoding Mucin protein, that are associated with gut permeability. | 6 weeks
  Genetic variants such as MUC2 will be determined where consent for genetic analysis is given.
Change in Systolic Blood Pressure (mmHg) | 6 weeks
  Change in Systolic Blood Pressure (mmHg) before and after the 6-week intervention.
Change in Diastolic Blood Pressure (mmHg) | 6 weeks
  Change in Diastolic Blood Pressure (mmHg) before and after the 6-week intervention.
Change in Heart Rate (beats/minute) | 6 weeks
  Change in Heart Rate (beats/minute) before and after the 6-week intervention.
Change in Waist-to-Hip Ratio | 6 weeks
  Change in Waist-to-Hip Ratio before and after the 6-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Noor K Al-Tameemi, PhD student candidate, Study Director — Nottingham Digestive Diseases Centre & NIHR Nottingham Biomedical Research Centre, Nottingham, University Hospitals NHS Trust and the University of Nottingham, Queens Medical Centre Nottingham, NG7 2UH; Guruprasad P Aithal, Professor, Principal Investigator — Nottingham Digestive Diseases Centre & NIHR Nottingham Biomedical Research Centre, Nottingham, University Hospitals NHS Trust and the University of Nottingham, Queens Medical Centre Nottingham, NG7 2UH; Jane Grove, Associate Professor, Study Director — Nottingham Digestive Diseases Centre & NIHR Nottingham Biomedical Research Centre, Nottingham, University Hospitals NHS Trust and the University of Nottingham, Queens Medical Centre Nottingham, NG7 2UH
Locations (3):
- United Kingdom (3):
  - Sir Peter Mansfield Imaging Centre, University of Nottingham, Nottingham
  - Nottingham Clinical Research Facility at Nottingham University Hospitals NHS Trust, Nottingham
  - University of Nottingham, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided